CLINICAL TRIAL: NCT02376036
Title: A Phase 1, First-in-Human, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of MGD010, a CD32B x CD79B Dual Affinity Re-Targeting (DART®) Bi-specific Antibody-Based Molecule, in Healthy Subjects
Brief Title: Phase 1 Study of MGD010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CP-MGD010-01
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Healthy Subjects
Keywords: Normal healthy volunteer
MeSH Terms: interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MGD010 (Experimental): Subjects will receive MGD010 through IV infusion.
  Interventions: Drug: MGD010
- Placebo (Placebo Comparator): Subjects will receive placebo through IV infusion.
  Interventions: Drug: Placebo
- MGD010 and HepA vaccine (Experimental): Subjects will receive MGD010 through IV infusion and HepA vaccine through an IM injection.
  Interventions: Drug: MGD010; Biological: Hepatitis A vaccine
- Placebo and HepA vaccine (Placebo Comparator): Subjects will receive placebo through IV infusion and HepA vaccine through an IM injection.
  Interventions: Drug: Placebo; Biological: Hepatitis A vaccine

INTERVENTIONS:
Drug: MGD010 — MGD010 is a CD32B x CD79B bi-specific antibody-based molecular construct referred to as a Dual Affinity Re-Targeting (DART) molecule. MGD010 will be administered as a single agent.
  Arms: MGD010; MGD010 and HepA vaccine
Drug: Placebo — Placebo comparator.
  Arms: Placebo; Placebo and HepA vaccine
Biological: Hepatitis A vaccine — Hepatitis A vaccine, inactivated
  Other Names: Vaqta
  Arms: MGD010 and HepA vaccine; Placebo and HepA vaccine

SUMMARY:
The primary goal of this Phase 1 study is to assess the safety and tolerability of one MGD010 intravenous (IV) infusion in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safety, tolerability and PK of MGD010, a CD32B x CD79B DART bi-specific antibody-based molecule. This study will be conducted as a double-blind, randomized, placebo controlled, single ascending dose study among healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years of age
* Body mass index (BMI) of 18 to 30 kg/m2, inclusive

Exclusion Criteria:

* Women of child-bearing potential;
* Women who are pregnant or breast-feeding
* Any significant acute or chronic medical illness
* Any major surgery within 4 weeks of study drug administration
* Active or latent tuberculosis (TB)
* Active or latent Hepatitis B, Hepatitis C or HIV infection
* History of allergy to monoclonal antibodies, any significant drug allergy (such as anaphylaxis), or hypersensitivity to any components of the test or reference investigational product formulation.
* Evidence of organ dysfunction or any clinically significant deviation from normal
* Vaccination with any live vaccine, or use of any prescription drugs, within 4 weeks of study drug administration
* Known history of infection or exposure to Hepatitis A virus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as assessed by AEs and SAEs | up to Day 57

SECONDARY OUTCOMES:
Serum concentration (pharmacokinetics) of MGD010 | up to Day 57
Incidence of MGD010 anti-drug antibodies (ADA) | up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (1):
- PAREXEL Baltimore Early Phase Clinical Unit, Baltimore, Maryland, United States